CLINICAL TRIAL: NCT06788392
Title: The Effect of Reminiscence Therapy Applied to Elderly Individuals Staying in Nursing Homes on Constipation and General Comfort
Brief Title: Nursing Homes on Constipation and General Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun Huzurevi Yaşlı Bakım ve Rehabilitasyon Merkezi (Other Government)
Collaborators: Kafkas University (Other)
Responsible Party: Principal Investigator, KEVSER KASAP, Nurse, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-KK-01; Kevser KASAP (Other: Giresun Nursıng Home Elderly Care And Rehabılıtatıon Center)
Record Dates: First submitted 2024-12-02; First posted 2025-01-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Constipation; Nursing Caries
Keywords: the elderly; constipation; comfort; reminiscence therapy
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Block randomisation will be used to ensure that the number of patients in each group is balanced. Patients will be divided into two groups, each group consisting of at least 38 people, by a statistician who is not involved in the study, using a table of random numbers.
Who Masked: Outcomes Assessor
Masking Description: In the study, blinding will be performed only in the assignment-randomisation to groups and statistical analysis of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Experimental): Group receiving reminiscence therapy 2 days a week
  Interventions: Other: reminiscence therapy
- control (No Intervention): The group in which no intervention and receiving routine nursing care

INTERVENTIONS:
Other: reminiscence therapy — Reminiscence Therapy is a supportive care model that has been used in recent years and increases life comfort.
  Arms: interventional

SUMMARY:
The Effect of Reminiscence Therapy on Constipation Applied to Elderly Individuals Staying in a Nursing Home in Giresun Province

DETAILED DESCRIPTION:
Research; This study will be conducted to determine the effect of reminiscence therapy, given once or twice a week to elderly people living in nursing homes, on constipation by reducing stress levels. It is thought that the results obtained will provide evidence for reducing constipation, which significantly limits life. Patients who complain of constipation at the Nursing Home Elderly Care and Rehabilitation Center, who voluntarily agree to participate in the research and who meet the sample selection criteria will be included in the study. Patient information will be collected and the research pre-test, post-test and application will be carried out face to face.

ELIGIBILITY:
Inclusion criteria for the study:

* Those aged 65 and over,
* Able to answer all questions and be communicative,
* Scoring 24 or above from the Mini Mental test,
* Agreeing to participate in the research,
* Diagnosed with constipation by the institution physician and meeting the Rome III Constipation Diagnostic Criteria,
* There is no deterioration in skin integrity or infection in the abdominal area,
* No diarrhea,
* Individuals without a history of abdominal surgery will be included in the study.

Exclusion Criteria

* Psychiatric drug users,
* Those who score below 24 on the Mini Mental Test,
* Those who do not meet the Rome III Diagnostic Criteria for Constipation,
* Those with impaired skin integrity or infection in the abdominal area,
* People with diarrhoea,
* History of abdominal surgery Those who refused to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Constipation Severity Scale (CSS) General Comfort | Constipation levels will be measured at the begining of the study (pre-test) and end of the intervention of the 5 weeks (post test)
  It was developed by Varma et al. in 2008. It is a scale for determining the frequency, intensity and difficulty/difficulty during defecation.
Defecation Monitoring Form in a Standard Diary (DMFSD) | Constipation status will be monitored at the beginning of the study and daily for 5 weeks
  In the form developed by Pamuk et al. (2003) there is a 7-day follow-up schedule consisting of 5 items, including the number of defecation, the amount of stool, the stool consistency, the feeling of buckling during defecation and the feeling of not fully emptying after defecation. For each symptom of constipation, all scores collected during the pre-treatment (7 days), sequence of application (21 days) and post-treatment (7 days) days were calculated by dividing the number of defecations performed within the same days.
General Comfort Questionnaire | Comfort levels will be measured at the begining of the study (pre-test) and end of the intervention of the 5 weeks (post test)
  It was developed by Kolcaba in 1992. A validity and reliability study was conducted by Kuğuoğlu and Karabacak in 2004. The General Comfort Scale is used to determine the comfort needs and to evaluate the state of achieving the result of increasing the expected comfort with the nursing interventions that constitute comfort, which includes three levels (relief, relaxation and superiority) and four dimensions (physical, psychospiritual, sociocultural and environmental) that constitute the theoretical factors of comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun Huzurevi Yaşli Bakim Ve Rehabilitasyon Merkezi, Giresun, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is the request of the individuals who participated in my study.